CLINICAL TRIAL: NCT03290339
Title: Preliminary Study About the Feasibility of Ambulatory Hysterectomy: Bicentric Study in Caen UH and Amiens UH
Brief Title: Feasibility of Ambulatory Hysterectomy
Acronym: AMETHYST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: Amiens University Hospital (Other)
Responsible Party: Principal Investigator, Raffaele FAUVET, professor, University Hospital, Caen
Other Study IDs: 2017-A01505-48
Record Dates: First submitted 2017-09-18; First posted 2017-09-21 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Surgery; Maternal, Uterus or Pelvic Organs, Affecting Fetus
Keywords: one-day surgery; hysterectomy; ambulatory
MeSH Terms: interventions — Hysterectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: hysterectomy — laparoscopic hysterectomy and vaginal hysterectomy

SUMMARY:
Hysterectomy is one of the most performed surgery in women. Public authorities wish that one-day surgery become a majority and hysterectomy could be part of it in the future. The aim of this study is to determine the feasibility of ambulatory hysterectomy.

Patients and methods: Investigators will realize an observational descriptive survey based on questionnaires in two surgical gynecology units. Women under 70 years old, who undergo hysterectomy will be included.

ELIGIBILITY:
Inclusion Criteria:

* women, undergo surgery for hysterectomy by laparoscopy or vaginal procedure

Exclusion Criteria:

* comorbidities included: heart disease, anti-coagulant treatment, anti-aggregant treatment; sleep apnea syndrome, laparotomy laparoconversion if hysterectomy associated with appendectomy and/or, omentectomy and/or, lymph nodes dissection

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women more than 18 and Under 70 years old who undergo hysterectomy by laparoscopy or vaginal procedure in one the two units
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-09-06 (Actual); Primary Completion 2019-09-06 (Estimated); Study Completion 2019-12-06 (Estimated)

PRIMARY OUTCOMES:
PADSS score | Day 0 post surgery

SECONDARY OUTCOMES:
patient satisfaction | Day 1
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: raffaele Fauvet, MD, PhD, Principal Investigator — Caen UH
Locations (1):
- Caen university hospital, Caen, Calvados, France

IPD SHARING:
Plan to Share IPD: No